CLINICAL TRIAL: NCT02741271
Title: A Phase III, Randomized, Active-Controlled, Parallel-Group Clinical Trial to Study the Efficacy and Long-Term Safety of Mometasone Furoate/Formoterol Fumarate (MF/F, MK-0887A [SCH418131]), Compared With Mometasone Furoate (MF, MK-0887 [SCH032088]), in Children With Persistent Asthma
Brief Title: Study of Efficacy and Long-Term Safety of Mometasone Furoate in Combination With Formoterol Fumarate Versus Mometasone Furoate in Children (5 to 11 Years of Age) With Persistent Asthma (MK-0887A-087)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0887A-087; MK-0887A-087 (Other: Merck Registration Number); 2009-010110-30 (EudraCT Number)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BID protein, human; Albuterol; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: 1:1 randomization to double-blinded MF/F MDI 100/10 mcg BID and MF MDI 100 mcg BID
Oversight: Data Monitoring Committee: No

ARMS (2):
- MF/F MDI 100/10 mcg BID (Experimental): Eligible participants will be assigned randomly to receive double-blinded MF/F MDI 100/10 mcg BID for 24 weeks.
  Interventions: Drug: MF MDI 100 mcg BID (Open Label); Drug: MF/F MDI 100/10 mcg BID; Drug: Albuterol/Salbutamol PRN; Drug: Prednisone/Prednisolone
- MF MDI 100 mcg BID (Active Comparator): Eligible participants will be assigned randomly to receive double-blinded MF MDI 100 mcg BID for 24 weeks.
  Interventions: Drug: MF MDI 100 mcg BID (Open Label); Drug: MF MDI 100 mcg BID; Drug: Albuterol/Salbutamol PRN; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: MF MDI 100 mcg BID (Open Label) — Eligible participants will receive open-label MF MDI 100 mcg BID during a 2-week run-in period.
  Other Names: ASMANEX HFA®; SCH 032088 (MK-0887)
Drug: MF/F MDI 100/10 mcg BID — After a 2 week run-in on open-label MF MDI 100 mcg BID, eligible participants will receive double-blinded treatment with MF/F MDI 100/10 mcg BID.
  Other Names: DULERA®/ZENHALE®; SCH 418131 (MK-0887A)
  Arms: MF/F MDI 100/10 mcg BID
Drug: MF MDI 100 mcg BID — After a 2 week run-in on open-label MF MDI 100 mcg BID, eligible participants will receive double-blinded treatment with MF MDI 100 mcg BID.
  Other Names: ASMANEX HFA®; SCH 032088 (MK-0887)
  Arms: MF MDI 100 mcg BID
Drug: Albuterol/Salbutamol PRN — Participants may use study-provided short-acting beta agonist (SABA), albuterol/salbutamol, as needed (PRN) for the relief of asthma symptoms.
Drug: Prednisone/Prednisolone — Participants may use a systemic corticosteroid (prednisone/prednisolone) for acute asthma worsening per investigator discretion.

SUMMARY:
This study compares the 12-week efficacy and 24-week safety of mometasone furoate/formoterol fumarate (MF/F) 100/10 mcg and mometasone furate (MF) 100 mcg, both administered twice daily (BID) via metered-dose inhaler (MDI) in children aged 5 to 11 years with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of asthma of ≥ 6-months duration according to the Global Initiative for Asthma (GINA) guidelines
* Has asthma that is adequately controlled on a stable dose of inhaled corticosteroid (ICS) combined with long-acting beta-agonist (LABA) ≥ 4 weeks
* Is able to demonstrate an FEV1 >60% and ≤90% predicted
* Is able to demonstrate an increase in absolute FEV1 of at least 12% within 30 minutes after administration of albuterol/salbutamol.
* Is able to use an MDI (without spacer), use a peak flow meter, and perform spirometry correctly.
* Is willing (with consent of their parent(s)/guardian) to discontinue previously prescribed asthma medication, if there is no inherent harm in changing the participant's current asthma therapy.
* Has laboratory tests that are clinically acceptable to the investigator.

Exclusion Criteria:

* Requires >8 inhalations per day of albuterol (100 mcg per actuation), and/or >2 nebulized treatments per day of 2.5 mg albuterol on any 2 consecutive days
* Has a clinical worsening of asthma that results in emergency room visit (for an asthma exacerbation), hospitalization due to asthma, or treatment with additional, excluded asthma medication (other than SABA) between the Screening and Baseline visits.
* Is considered by the investigator to have unstable asthma at the end of the run-in period
* Has had > 4 asthma exacerbations (defined as a worsening of asthma requiring systemic corticosteroid use and/or ≥ 24-hour stay in an emergency department, urgent care center, or hospital) within 1 year prior to visit 1
* Has had a history of life-threatening asthma
* Has a clinically significant condition or situation, other than the condition being studied which may interfere with trial evaluations, participant safety, or optimal participation in the trial

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weinstein CLJ, Gates D, Zhang X, Varnell T, Mok W, Vermeulen JH, Amar NJ, Jain N. A phase 3 study evaluating the safety and efficacy of a pediatric dose of mometasone furoate with and without formoterol for persistent asthma. Pediatr Pulmonol. 2020 Apr;55(4):882-889. doi: 10.1002/ppul.24667. Epub 2020 Feb 5. PMID 32022483

RESULTS

PARTICIPANT FLOW:
Groups:
- MF/F MDI 100/10 mcg BID: MF/F administered by MDI, given as 100/10 mcg BID
- MF MDI 100 mcg BID: MF administered by MDI, given as 100 mcg BID
Period: Overall Study
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Started | 91 | 90
Completed | 89 | 88
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.7) | 9.1 (1.7) | 9.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 89
  Male | 45 | 47 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 38 | 78
  Not Hispanic or Latino | 51 | 52 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 43 | 41 | 84
  More than one race | 33 | 37 | 70
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning (AM) Post-Dose % Predicted Forced Expiratory Volume in One Second (FEV1) in the Area Under the Curve (AUC)0-60
Description: This endpoint reflects changes in lung function data (forced expiratory volume in 1 second) measured across 0 to 60 minutes post-dose (at 0, 5, 15, 30 and 60 minutes) and averaged across study visits in the Treatment Period (Day 1, Week 1, Week 4, Week 8 and Week 12) compared to Baseline. Baseline was the average of % predicted FEV1 values at 30 min and 0 min pre-dose. At each visit, the area under the curve is calculated over the post-dose timepoints. Units are standardized to percent predicted FEV1 by dividing the AUC calculation by the duration of the observed AUC.
Time Frame: Baseline, and average of Day 1, Weeks 1, 4, 8, and 12
Population: All participants who received at least one dose of randomized trial medication with at least one primary efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Percent predicted FEV1
  Baseline | 79.21 (11.44) | 78.48 (12.79)
  Change from Baseline | 8.99 (8.29) | 3.96 (5.92)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method, using the constrained Longitudinal Data Analysis (cLDA) model for missing data; LSM Difference = 5.21, 95% CI 2-sided [3.21 to 7.20] — Between-Treatment Difference

2. Primary Outcome: Count (Percentage) of Participants Experiencing At Least One Adverse Event (AE)
Description: An Adverse Event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 26 weeks
Population: All randomized participants who received at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Groups:
- Total: All treated participants
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | Total
Number analyzed (Participants) | 91 | 90 | 181
Participants | 37 | 52 | 89

3. Primary Outcome: Count (Percentage) of Participants Discontinuing From Study Medication Due to An AE
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of trial medication
Measure: Count of Participants; unit: Participants
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | Total
Number analyzed (Participants) | 91 | 90 | 181
Participants | 0 | 3 | 3

4. Secondary Outcome: Change From Baseline AM Post-Dose Percent Predicted FEV1 on Day 1 of Treatment
Description: The key secondary objective was to determine the onset of action for the efficacy of MF/F MDI 100/10 mcg BID, compared with MF MDI 100 mcg BID. The post-dose AM % predicted FEV1 was averaged sequentially, and the change from baseline on Day 1 was assessed. This key secondary endpoint was controlled for multiplicity in a step-down fashion, based on trial success defined as a statistically significant improvement in the primary endpoint for MF/F vs MF. Missing data were imputed using control-based multiple imputations with the cLDA model.
Time Frame: Baseline and Day 1, measured at 4 hr, 2 hr and 60, 30, 15, and 5 min, post-dose time points
Population: All participants who received at least one dose of randomized trial medication with at least one efficacy evaluation
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Percent predicted FEV1
  Baseline | 79.21 (11.44) | 78.48 (12.79)
  Change from Baseline (4 hr post-dose on Day 1) | 11.61 (10.31) | 5.68 (7.38)
  Change from Baseline (2 hr post-dose on Day 1) | 12.71 (9.53) | 5.87 (6.52)
  Change from Baseline (60 min post-dose on Day 1) | 11.05 (8.51) | 4.92 (6.06)
  Change from Baseline (30 min post-dose on Day 1) | 9.56 (7.02) | 3.05 (4.99)
  Change from Baseline (15 min post-dose on Day 1) | 8.00 (7.12) | 1.38 (4.42)
  Change from Baseline (5 min post-dose on Day 1) | 5.20 (6.93) | 0.95 (4.33)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 6.05, 95% CI 2-sided [3.53 to 8.56] — Between-Treatment Difference at 4 hr Post-Dose
Statistical Analysis 2: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 7.04, 95% CI 2-sided [4.74 to 9.35] — Between-Treatment Difference at 2 hr Post-Dose
Statistical Analysis 3: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 6.19, 95% CI 2-sided [4.09 to 8.28] — Between-Treatment Difference at 60 min Post-Dose
Statistical Analysis 4: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 6.89, 95% CI 2-sided [5.10 to 8.67] — Between-Treatment Difference at 30 min Post-Dose
Statistical Analysis 5: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 6.64, 95% CI 2-sided [4.89 to 8.39] — Between-Treatment Difference at 15 min Post-Dose
Statistical Analysis 6: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA with multiple imputation; Primary Analysis Method; LSM Difference = 4.20, 95% CI 2-sided [2.50 to 5.91] — Between-Treatment Difference at 5 min Post-Dose

5. Secondary Outcome: Change From Baseline AM Post-Dose % Predicted FEV1 AUC 0-4 Hours on Day 1 and Week 12 of Treatment
Description: This endpoint reflects changes in lung function data (forced expiratory volume in 1 second) measured across 0 to 4 hours post-dose on Day 1 and Week 12 compared to Baseline. Baseline was the average of 30 and 0 minutes pre-dose % predicted FEV1 values. The AUC was calculated over the scheduled timepoints of 0 min, 5 min, 15 min, 30 min, 60 min, 2 hr and 4 hr post-dose. Units are standardized to percent predicted FEV1 by dividing the AUC calculation by the duration of the observed AUC.
Time Frame: Baseline, Day 1 and Week 12
Population: All participants who received at least one dose of randomized trial medication with at least one efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 89
Percent predicted FEV1
  Baseline | 79.21 (11.44) | 78.48 (12.79)
  Change from Baseline on Day 1 | 7.13 (5.35) | 2.70 (3.09)
  Change from Baseline at Week 12 | 7.56 (11.20) | 4.87 (7.72)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p < 0.001, cLDA; Secondary Outcome Measure on Day 1; LSM Difference = 6.32, 95% CI 2-sided [4.36 to 8.27] — Between-Treatment Difference at 4 hr Post-Dose
Statistical Analysis 2: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p = 0.026, cLDA; Secondary Outcome Measure at Week 12; LSM Difference = 3.33, 95% CI 2-sided [0.41 to 6.26] — Between-Treatment Difference at 4 hr Post-Dose

6. Secondary Outcome: Change From Baseline in AM Pre-Dose % Predicted FEV1 With MF/F MDI 100/10 mcg BID or MF MDI 100 mcg BID Over the First 12 Weeks of Treatment
Description: The change from baseline in AM pre-dose % predicted FEV1 with MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID averaged over 12 weeks treatment was assessed. This secondary analysis of the change from baseline used the cLDA method without multiple imputation. A model-based MAR approach was used for missing data.
Time Frame: Baseline and Weeks 4, 8, and 12 (Averaged)
Population: All participants who received at least one dose of randomized trial medication with at least one efficacy evaluation across the treatment period.
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Percent predicted FEV1
  Baseline | 79.21 (11.44) | 78.22 (12.93)
  Change from Baseline (Weeks 4, 8, and 12) | 1.51 (7.15) | 0.44 (5.49)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority; p = 0.197, cLDA; Secondary Outcome Measure; LSM Difference = 1.63, 95% CI 2-sided [-0.85 to 4.11] — Between-Treatment Difference

7. Secondary Outcome: Mean Change From Baseline in Total Daily Use of Short-Acting Beta-Agonist (SABA) Rescue Medication With MF/F MDI 100/10 mcg BID or MF MDI 100 mcg BID Over the First 12 Weeks of Treatment
Description: To evaluate the efficacy of MF/F MDI 100/10 mcg BID compared with MF MDI 100 mcg BID, the change from baseline in total daily short-acting beta-agonist (SABA) use (puffs per day) was averaged and assessed. All participants received SABA MDIs (albuterol 90 mcg or salbutamol 100 mcg) for as-needed relief of asthma symptoms. This secondary analysis of the change from baseline used the cLDA method without multiple imputation.A model-based MAR approach was used for missing data.
Time Frame: Baseline and Weeks 1-12 (Averaged)
Population: All participants who received at least one dose of randomized trial medication with at least one efficacy evaluation
Measure: Mean (Standard Deviation); unit: Puffs per day
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Puffs per day
  Baseline | 0.25 (0.66) | 0.13 (0.50)
  Change from Baseline Over Weeks 1-12 (Average) | -0.12 (0.58) | -0.02 (0.52)

8. Secondary Outcome: Participants Using SABA Rescue Medication Across Weeks 1-12 of the Treatment Period
Description: To evaluate the efficacy of MF/F MDI 100/10 mcg BID compared with MF MDI 100 mcg BID, the number of participants using SABA rescue medication in Weeks 1-12 (individually) of the double-blind treatment period was assessed. All participants received SABA MDIs (albuterol 90 mcg or salbutamol 100 mcg) for as-needed relief of asthma symptoms.
Time Frame: Baseline and Weeks 1-12 (Averaged)
Population: Data were provided for all participants who received at least one dose of randomized trial medication and had at least one efficacy evaluation.
Measure: Number; unit: Participants
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Participants
  Baseline | 23 | 17
  Weeks 1-12 | 41 | 45

9. Secondary Outcome: Participants Whose SABA Rescue Medication Use Increased Across Weeks 1-12 of the Treatment Period
Description: To evaluate the efficacy of MF/F MDI 100/10 mcg BID compared with MF MDI 100 mcg BID, the number of participants whose use of SABA rescue medication increased in Weeks 1-12 (individually) of the double-blind treatment period was assessed. All participants received SABA MDIs (albuterol 90 mcg or salbutamol 100 mcg) for relief of asthma symptoms.
Time Frame: Weeks 1-12 (Averaged)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
Number analyzed (Participants) | 91 | 90
Participants | 24 | 34

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve of Mometasone Furoate From Time 0 to 12 Hours (AUC0-12)
Description: Blood samples were collected predose, and 0.75, 1.5, 3, 8, and 12 hours postdose at Week 12 in a subset of participants who consented to take part in a PK sub-trial. Per protocol, descriptive MF pharmacokinetics were summarized without regard to treatment assignment.
Time Frame: Predose, 0.75, 1.5, 3, 8, and 12 hours postdose at Week 12
Population: Participants who consented to take part in the PK sub-trial and had evaluable data for AUC(0-12).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Groups:
- Pooled MF/F 100/10 mcg and MF 100 mcg: MF/F 100/10 mcg BID or MF 100 mcg BID, administered by MDI
Arm/Group | Pooled MF/F 100/10 mcg and MF 100 mcg
Number analyzed (Participants) | 10
hr*pg/mL | 109 (55.8)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve of Mometasone Furoate From Time 0 to Time of Last Measurable Concentration (AUC0-last)
Description: as for outcome 10
Time Frame: Predose, 0.75, 1.5, 3, 8, and 12 hours postdose at Week 12
Population: Participants who consented to take part in the PK sub-trial and had evaluable data for AUC(0-last).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Pooled MF/F 100/10 mcg and MF 100 mcg
Number analyzed (Participants) | 11
hr*pg/mL | 106 (53.5)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Mometsone Furoate
Description: as for outcome 10
Time Frame: Predose, 0.75, 1.5, 3, 8, and 12 hours postdose at Week 12
Population: Participants who consented to take part in the PK sub-trial and had evaluable data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Pooled MF/F 100/10 mcg and MF 100 mcg
Number analyzed (Participants) | 11
pg/mL | 16 (68.2)

13. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Mometsone Furoate
Description: as for outcome 10
Time Frame: Predose, 0.75, 1.5, 3, 8, and 12 hours postdose at Week 12
Population: Participants who consented to take part in the PK sub-trial and had evaluable data for Tmax.
Measure: Median (Full Range); unit: hr
Arm/Group | Pooled MF/F 100/10 mcg and MF 100 mcg
Number analyzed (Participants) | 11
hr | 1.47 [0.50 to 12.00]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: All participants who received double-blind treatment
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90
Serious Adverse Events (participants affected / at risk) | 1/91 | 2/90
Other Adverse Events (participants affected / at risk) | 22/91 | 32/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 100/10 mcg BID (N=91) | MF MDI 100 mcg BID (N=90)
Epididymitis (Infections and infestations) | 0 | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 100/10 mcg BID (N=91) | MF MDI 100 mcg BID (N=90)
Influenza (Infections and infestations) | 5 (5) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (3) | 8 (9)
Pharyngitis (Infections and infestations) | 1 (1) | 6 (6)
Rhinitis (Infections and infestations) | 0 | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 14 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT02741271/Prot_SAP_000.pdf